CLINICAL TRIAL: NCT01314417
Title: Treatment of Non-infectious Panuveitis, Intermediate and Posterior Uveitis Associated Macular Edema With Intravitreal Methotrexate
Brief Title: Treatment of Non-infectious Intermediate and Posterior Uveitis Associated Macular Edema With Intravitreal Methotrexate
Acronym: MEXX
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: This study was terminated due to lack of recruitment.
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Nida Sen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110107; 11-EI-0107 (Other: NIH Office of Protocol Services)
Record Dates: First submitted 2011-03-11; First posted 2011-03-14 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2019-03-27 (Actual); Status verified 2018-07

CONDITIONS: Non-infectious Intermediate and Posterior Uveitis
Keywords: Uveitis; Macular Edema; Methotrexate
MeSH Terms: conditions — Uveitis, Posterior; Uveitis; Macular Edema | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate (Experimental): 400 μg/100 μL injection
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — 400 μg/100 μL monthly injections for the first 3 months, then as needed per the treatment criteria

SUMMARY:
BACKGROUND:

Uveitis comprises of a group of diseases associated with inflammation of the eye that can lead to vision loss. Some people with uveitis also have macular edema (swelling of the retina at the back of the eye). Uveitis and macular edema are treated with medications and sometimes surgery, but treatment does not always prevent vision loss. Previous research has shown that injections of methotrexate into the eye of people with eye disease other than uveitis can help relieve the inflammation, or swelling, that causes macular edema and can slow visual loss. However, it has not yet been approved as a treatment for macular edema associated with uveitis.

OBJECTIVES:

To evaluate the safety and effectiveness of methotrexate injections as a treatment for macular edema associated with uveitis.

ELIGIBILITY:

Individuals at least 18 years of age who have been diagnosed with uveitis and macular edema in at least one eye.

DESIGN:

* This study requires at least nine visits to the National Eye Institute study clinic over a period of 6 months (24 weeks).
* Participants will be screened with a physical and ophthalmic examination, medical history, blood and urine tests, and additional eye and other tests as needed.
* Participants will receive a methotrexate injection in a selected treatment eye. After the injection, participants will receive antibiotic eye drops to place in the eye three times a day for the 3 days following the injection, leucovorin (folic acid) drops to place in the eye four times a day for 1 week following the injection, and a dose of folic acid to be taken by mouth the day after the injection.
* Participants who tolerate the initial injection may continue to receive injections in their study eye every month for 6 months. After 6 months, participants who show improvement from the injections may be evaluated to receive additional injections every 4 to 8 weeks until researchers end the study.

DETAILED DESCRIPTION:
OBJECTIVE:

The study objective is to investigate the safety, tolerability and potential efficacy of intravitreal injections of methotrexate as a possible treatment for chronic macular edema secondary to panuveitis, posterior or intermediate uveitis.

STUDY POPULATION:

Five participants with chronic macular edema associated with panuveitis, posterior or intermediate uveitis will be initially enrolled. However, up to an additional two participants may be enrolled to account for participants who withdraw from the study prior to reaching Week 12. Eligibility criteria include macular edema in the study eye, which has not been responsive to conventional immunosuppressive therapy in the past three months, or the participant experienced a recurrence of macular edema while on conventional immunosuppressive therapy.

STUDY DESIGN:

In this single-center, prospective, uncontrolled, unmasked, Phase I/II clinical trial, intravitreal injections of methotrexate at a dose of 400 μg per 100 μL will be administered. There will be an induction phase and a pro re nata (PRN) phase. During the induction phase, participants will receive injections at baseline and Weeks 4, 8, 12, 16 and 20 in their study eye unless contraindicated. Additional safety visits will occur at Weeks 1 and 2. Beginning at Week 24, participants who agree to remain in the study will undergo evaluation for injection in the study eye PRN every 4-8 weeks. These participants will be followed for 4-8 weeks after the last enrolled participant completes his/her Week 24 visit.

OUTCOME MEASURES:

The primary outcome is the number of participants who meet the definition of treatment success within 12 weeks from baseline. Treatment success is defined as achieving at least a 1-step decrease in the LogScore scale for central macular thickness. Secondary outcomes include changes in Early Treatment Diabetic Retinopathy Study (ETDRS) best-corrected visual acuity (BCVA), changes in excess retinal thickening, changes in macular thickness, changes in intraocular inflammation on clinical exam, changes in leakage as seen on fluorescein angiography (FA), changes in autofluorescence patterns seen on fundus autofluorescence (FAF) imaging and observation of dose reductions of systemic immunosuppression or steroids. Safety outcomes include the number and severity of adverse events, systemic and ocular toxicities, electrophysiologic changes assessed by full-field electroretinography (ERG) and number of withdrawals.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Participant must be 18 years of age or older.
2. Participant must understand and sign the protocol's informed consent document.
3. Participant is willing to comply with the study procedures and return for all study visits.
4. Participant has chronic macular edema secondary to non-infectious panuveitis, posterior or intermediate uveitis in at least one eye (the study eye) that has:

   1. not been responsive to conventional immunosuppressive therapy in the past 3 months; OR
   2. recurred while on conventional immunosuppressive therapy.
5. Participant has central macular thickness of ≥ 270 microns in the study eye.
6. Participant has visual acuity of 20/400 or better (≥ 19 ETDRS letters) in the study eye.
7. Female participants of childbearing potential must not be pregnant or breast-feeding, must have a negative serum pregnancy test at screening and must be willing to undergo serum pregnancy tests throughout the study.
8. Both female participants of childbearing potential (see Appendix 1 for definition) and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two acceptable methods of contraception throughout the course of the study and for six months after the last study medication injection. Acceptable methods of contraception include:

   * hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
   * intrauterine device,
   * barrier methods (diaphragm, condom) with spermicide, or
   * surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

1. Participant is in another investigational study and actively receiving investigational therapy for macular edema.
2. Participant has evidence of infectious panuveitis, posterior or intermediate uveitis in either eye.
3. Participant is expected to need ocular surgery in the study eye during the course of the trial.
4. Participant had intraocular surgery in the study eye within the past 90 days.
5. Participant had an injection of bevacizumab or ranibizumab within the past four weeks in the study eye.
6. Participant had an injection of triamcinolone within the past six weeks in the study eye.
7. Participant has a systemic condition that, in the opinion of the investigator, would preclude participation in the study.
8. Participant has significant cataract or media opacity in the study eye that makes posterior segment visualization difficult as determined by investigator.
9. Participant has a confirmed positive serologic and/or molecular test for HIV-1/2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-02; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Lardenoye CW, van Kooij B, Rothova A. Impact of macular edema on visual acuity in uveitis. Ophthalmology. 2006 Aug;113(8):1446-9. doi: 10.1016/j.ophtha.2006.03.027. PMID 16877081
- [Background] Kiss CG, Barisani-Asenbauer T, Maca S, Richter-Mueksch S, Radner W. Reading performance of patients with uveitis-associated cystoid macular edema. Am J Ophthalmol. 2006 Oct;142(4):620-4. doi: 10.1016/j.ajo.2006.05.001. PMID 17011854
- [Background] Rothova A. Inflammatory cystoid macular edema. Curr Opin Ophthalmol. 2007 Nov;18(6):487-92. doi: 10.1097/ICU.0b013e3282f03d2e. PMID 18163001
- [Background] van Kooij B, Rothova A, de Vries P. The pros and cons of intravitreal triamcinolone injections for uveitis and inflammatory cystoid macular edema. Ocul Immunol Inflamm. 2006 Apr;14(2):73-85. doi: 10.1080/09273940500545684. PMID 16597536
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2011-EI-0107.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate: Participants will receive an intravitreal injection of 400 μg per 100 μL of methotrexate at baseline and Weeks 4 and 8, then as needed per the treatment criteria.
Period: Overall Study
Arm/Group | Methotrexate
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.0 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Meet the Definition of Treatment Success Within 12 Weeks From Baseline.
Description: Treatment success is defined as achieving at least a 1-step decrease in the LogScore scale for central macular thickness.
  A decrease of at least 1-step on the logOCT scale, where Change in logOCT=log(follow-up thickness/200) - log(baseline thickness/200) is considered clinically significant. A 1-step decrease is equivalent to at least a 20% improvement of central macular thickness and represents greater than twice the variability of retinal thickness measurements (approximately 25-30 µ).
  Examples of OCT measurements with their corresponding LogScore, where LogScore=10xlogOCT are as follows:
  LogScore 0 = OCT 200 µm, LogScore 1 = OCT 250 µm, LogScore 2 = OCT 320 µm, LogScore 3 = OCT 400 µm, LogScore 4 = OCT 500 µm, LogScore 5 = OCT 640 µm, LogScore 6 = OCT 800 µm, LogScore 7 = OCT 1000 µm
Time Frame: 12 weeks
Measure: Number; unit: Participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Participants | 2

2. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 4 Weeks Compared to Baseline
Description: Excess retinal thickening was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria.
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 7.2 (2.3)

3. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 8 Weeks Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 9.9 (2.3)

4. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 12 Weeks Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 6.1 (6.6)

5. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 16 Weeks Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 16
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 13.6 (9.3)

6. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 20 Weeks Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 4.9 (4.4)

7. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Excess Retinal Thickening in the Study Eye at 24 Weeks Compared to Baseline
Description: as for outcome 2
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
percentage of change from baseline | 10.6 (10.3)

8. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 4 Weeks Compared to Baseline
Description: Central-subfield macular thickness was assessed by spectral-domain optical coherence tomography (Cirrus HD-OCT; Carl Zeiss Meditec, Dublin, CA), a non-invasive imaging technique that uses long-wavelength light to capture micrometer-resolution cross-sectional images from biological tissue.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria.
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 60.5 (44.5)

9. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 8 Weeks Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 72.0 (19.8)

10. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 12 Weeks Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 99.0 (63.6)

11. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 16 Weeks Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 16
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 87.5 (20.5)

12. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 20 Weeks Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 46.0 (52.3)

13. Secondary Outcome: Change in Optical Coherence Tomography (OCT) Central Macular Thickness in the Study Eye at 24 Weeks Compared to Baseline
Description: as for outcome 8
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: µm
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
µm | 101.0 (118.8)

14. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 4 Weeks Compared to Baseline
Description: Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria.
Time Frame: Baseline and Week 4
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
ETDRS Letters | 6.0 (4.2)

15. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 8 Weeks Compared to Baseline
Description: as for outcome 14
Time Frame: Baseline and Week 8
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
ETDRS Letters | 1.5 (2.1)

16. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 12 Weeks Compared to Baseline
Description: as for outcome 14
Time Frame: Baseline and Week 12
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
ETDRS Letters | 3 (0)

17. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 16 Weeks Compared to Baseline
Description: as for outcome 14
Time Frame: Baseline and Week 16
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
ETDRS Letters | 1.5 (7.8)

18. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 24 Weeks Compared to Baseline
Description: as for outcome 14
Time Frame: Baseline and Week 24
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
ETDRS Letters | 1.5 (4.9)

19. Secondary Outcome: Changes in Early Treatment Diabetic Retinopathy Study (ETDRS) Best-corrected Visual Acuity (BCVA) in the Study Eye at 20 Weeks Compared to Baseline
Description: as for outcome 14
Time Frame: Baseline and Week 20
Measure: Mean (Standard Deviation); unit: ETDRS Letters
Units Other Than Participants: Eyes
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
Number analyzed (Eyes) | 2
ETDRS Letters | 1.5 (0.7)

20. Secondary Outcome: Number of Participants Presenting No Change in the Area of Leakage in the Study Eye as Seen on Fluorescein Angiography (FA) Imaging at Week 12 as Compared to Baseline
Description: Fluorescein angiography (FA) images were obtained via a standard digital imaging system (OIS, Sacramento, CA). Three retinal specialists independently graded the area of late fluorescein leakage (at approximately 10 minutes) in each eye using a region-of-interest tool in an image analysis software package (NIH ImageJ, Bethesda, MD).
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria.
Time Frame: Baseline and Week 12
Measure: Number; unit: participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
participants | 2

21. Secondary Outcome: Number of Participants Presenting No Change in the Area of Leakage in the Study Eye as Seen on Fluorescein Angiography (FA) Imaging at Week 24 as Compared to Baseline
Description: as for outcome 20
Time Frame: Baseline and Week 24
Measure: Number; unit: participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
participants | 2

22. Secondary Outcome: Number of Participants Presenting the Same Autofluorescence Patterns in the Study Eye as Seen on Fundus Autofluorescence (FAF) Imaging at Week 12 as Observed at Baseline
Description: Fundus autofluorescence patterns were assessed using fundus autofluorescence (FAF) imaging, a non-invasive technique that uses a confocal scanning ophthalmoscope to detect naturally-fluorescing lipofuscin.
  The participant's eye that met the study eye eligibility criteria was selected as the study eye. For cases in which both eyes met the study eye eligibility criteria, the study eye was selected according to the "choice of study eye in cases of bilateral disease" selection criteria outlined in the eligibility criteria.
Time Frame: Baseline and Week 12
Measure: Number; unit: participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
participants | 2

23. Secondary Outcome: Number of Participants Presenting the Same Autofluorescence Patterns in the Study Eye as Seen on Fundus Autofluorescence (FAF) Imaging at Week 24 as Observed at Baseline
Description: as for outcome 22
Time Frame: Baseline and Week 24
Measure: Number; unit: participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
participants | 2

24. Secondary Outcome: Number of Participants Experiencing a Complete Resolution of Fluid as Seen on OCT at Any Time During the Study Period
Time Frame: Baseline and Week 74
Measure: Number; unit: participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 2
participants | 0

25. Secondary Outcome: Observation of Dose Reduction of Systemic Immunosuppression or Steroids Over the Course of the Study Period
Description: This study terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and Week 74
Population: As this study terminated early due to lack of recruitment, data were not collected for this outcome.
Arm/Group | Methotrexate
Number analyzed (Participants) | 0

26. Secondary Outcome: Cytokine Analysis on Aqueous Samples to Assess Whether Intravitreal Injection of Methotrexate Affects Aqueous Inflammatory Cytokine Levels
Description: This study terminated early due to lack of recruitment; therefore, we chose not to report due to insufficient data.
Time Frame: Baseline and Week 74
Population: As this study terminated early due to lack of recruitment, data were not collected for this outcome.
Arm/Group | Methotrexate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Methotrexate
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Methotrexate (N=2)
Hypotony of eye (Eye disorders) | 1 (2)
Ear Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Staphylococcal skin infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Uveitis (Eye disorders) | 1 (1) — Worsening of uveitis in the non-study eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No